CLINICAL TRIAL: NCT05030961
Title: Implementation of a Team-based Virtual Clinic for Pediatric Cochlear Implants
Brief Title: Team-based Virtual Pediatric Cochlear Implant Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Stanley J. Glaser Foundation (Unknown)
Responsible Party: Principal Investigator, Chrisanda Sanchez, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20210584
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Cochlear Implant Candidate Group (Experimental): Participants who are in the process of receiving standard of care cochlear implant evaluation. Participants will receive a virtual team-based clinic as a part of the candidacy evaluation process for one year.
  Interventions: Behavioral: Virtual team-based clinic
- Established Cochlear Implant Recipient Group (Experimental): Participants who are established cochlear implant recipients. Participants will receive a virtual team-based clinic, including remote cochlear implant programming, for one year.
  Interventions: Behavioral: Virtual team-based clinic; Behavioral: Remote cochlear implant programming

INTERVENTIONS:
Behavioral: Virtual team-based clinic — Virtual team-based clinic will include consultation, counseling, and education from pediatric audiology, psychology, auditory verbal therapy, and education. Each session lasts approximately 30 minutes with a total of 3 sessions within the year.
Behavioral: Remote cochlear implant programming — Remote cochlear implant programming will be provided via Zoom on a study-provided encrypted laptop.
  Arms: Established Cochlear Implant Recipient Group

SUMMARY:
The purpose of this study is to see if remote visits for pediatric cochlear implant patients are possible. The investigator will be assessing whether a multi-disciplinary team approach can be achieved remotely for patients both undergoing the cochlear implant (CI) process and for those who have already been implanted.

ELIGIBILITY:
Inclusion Criteria:

New patients undergoing CI evaluation:

1. English speaking patients (parents can speak English and/or Spanish)
2. Ages 0-12 years who are cochlear implant candidates and undergoing the evaluation process

Established CI recipients:

1. English speaking patients (parents can speak English and/or Spanish)
2. Ages 1-12 with at least 6 months of CI experience with a company that has remote programming capacity

Exclusion Criteria:

1. Patients with families who speak languages other than English or Spanish
2. Patients who do not live in Florida
3. Patients who have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Electrode Impedances | Up to 1 year
  Electrode Impedances values, reported in kOhm, will be extracted from the cochlear implant software
Electrically evoked compound potential values | Up to 1 year
  Electrically evoked compound potential values, reported in mV, will be extracted from the cochlear implant software
Datalogging | Up to 1 year
  Datalogging, reported in hours per week, will be extracted from the cochlear implant software
Threshold/Upper stimulation levels | Up to 1 year
  As measured from the cochlear implant software
LittleEars questionnaire scores | Up to 1 year
  The LittleEars auditory questionnaire (LEAQ) uses parent responses to assess auditory behavior in children up to 24 months of age. The questionnaire is scored from 0 to 35 with 0 indicating poorer performance and 35 indicating better performance.
Auditory Skills Checklist (ASC) scores | Up to 1 year
  ASC has a Total Score ranges from zero to 70, with higher scores indicating development of increasingly complex listening skills

SECONDARY OUTCOMES:
Behavior Assessment System for Children version 3 (BASC-3) scores | Up to 1 year
  BASC-3 is scored 0-120 as a T score. Any scores between 60-70 is considered at risk / requires monitoring and scores greater than 70 are considered clinically significant / an area that likely requires therapeutic intervention.
Patient Health Questionnaire version 8 (PHQ-8) scores | Up to 1 year
  PHQ-8 has 8 items rated on a scale from "not at all" (0) to "nearly every day" (3), with higher scores indicating greater frequency of depressive symptoms. The sum of the items indicates the overall level of depressive symptoms indicating mild (5-9), moderate (10-14), moderately severe (15-19), and severe depressive symptoms (20- 24).
Generalized Anxiety Disorder version 7 (GAD-7) scores | Up to 1 year
  GAD-7 is a 7-item self-report questionnaire of anxiety symptomatology in the past 14 days. Respondents rate the frequency of each item during the past two weeks on a 0-3-point scale ranging from not at all (0) to nearly every day (3). The sum of the items indicates the overall level of anxiety symptoms indicating mild (0-4), moderate (5-9), moderately severe (10-14), and severe (15- 21).
Quality of Life- CI (QoL-CI) scores | Up to 1 year
  QoL-CI is scored 0-100 with higher scores indicating better quality of life.
Cochlear Implant Quality of Life-35 Profile (CIQOL-35 Profile) scores | Up to 1 year
  CIQOL-35 Profile is a 35 item questionnaire with a total score ranging from 0-100% with a higher score indicating a higher level of functional ability with a cochlear implant
Parenting Stress Index/Short Form (PSI) scores | Up to 1 year
  Parenting Stress Index/Short Form (PSI) contains 36 items rated on a 6-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree) and a total score. Higher scores indicate increased parenting stress.
Parenting Stress-CI scores | Up to 1 year
  Parenting Stress-CI is completed by the parent and scored from "not at all stressful" (0) to "very stressful" (3) with higher scores indicating greater degrees of parenting stress. For parents of children 0-5 years, there are 15 items. For parents of children 6-12 years there are 8 items.
Scale of Parental Involvement and Self-Efficacy-Revised (SPISE-R) scores | Up to 1 year
  The SPISE-R is comprised of 46 questions that uses a 7-point Likert scale to query parents' beliefs, knowledge, confidence, and actions relevant to supporting their child's auditory access and spoken language development. The total average score will range from 1 to 7 with 7 indicating the highest score / highest level of parental involvement and self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Chrisanda M Sanchez, AuD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No